CLINICAL TRIAL: NCT00297414
Title: An Analysis of Mortality in Subjects Who Participated in Three Studies of Galantamine in Mild Cognitive Impairment
Brief Title: An Observational Study for Analysis of Mortality in Participants Who Participated in Previous 3 Studies of Galantamine
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: SENIOR DIRECTOR, CLINICAL LEADER, Janssen R&D US
Other Study IDs: CR004240; GAL-COG-3002 (Other: Johnson & Johnson Pharmaceutical Research & Development, LLC)
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Dementia; Galantamine; Memory disorders; Isolated memory impairment; Alzheimer's disease
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Memory Disorders; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with mild cognitive impairment: Patients with mild cognitive impairment who were treated with galantamine or placebo in previous 3 clinical studies.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No study drug was administered to the patients. Data on vital status was obtained for patients with mild cognitive impairment who were treated with galantamine or placebo in previous 3 clinical studies.

SUMMARY:
The purpose of the study is to collect data of patients who were randomized (assignment of study medication by chance) and treated in 3 previous studies of galantamine (CR003145, CR002014 and CR005947) for the treatment of mild cognitive impairment (isolated memory impairment). This data were not recorded during the course of these 3 previous studies.

DETAILED DESCRIPTION:
The objective of this observational study is to ascertain follow-up vital status data for patients who were randomized (assignment of study medication by chance) and treated with galantamine or placebo in 3 previous studies (CR003145, CR002014 and CR005947). This study is designed to evaluate the imbalance of deaths that were initially recorded in the double-blind (neither physician nor patient knows the treatment that the patient receives) phases of two of these studies. Data will be combined from three sources: the databases of the 3 previous studies, forms from investigators, and data acquired during the present study. Investigator will obtain consent from the patients or their informant for participating in the study. Data on vital status will be obtained either from the patient or informant after obtaining informed consent. If a patient does not provide informed consent, documentation of contact with the patient will suffice as evidence that the patient is alive. If an informant does not provide informed consent or a patient cannot be contacted, medical or death records or death registers will be consulted when necessary to determine if a death occurred. If a patient was found to have died, the investigator records the cause of death, date of death, and the adverse events (unwanted consequence that occurs during the course of the clinical study, but not necessarily because of study medication) leading to death, by a review of medical records, autopsy records, and/or death certificates.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were randomized and treated with galantamine or placebo in 3 previous studies (CR003145, CR002014, and CR005947)

Exclusion Criteria:

* Patients not enrolled in above referenced studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population included patients randomized and treated with galantamine or placebo in 3 previous studies (CR003145, CR002014, and CR005947)
Sampling Method: Non-Probability Sample
Enrollment: 1083 (Actual)
Dates: Start 2004-06; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To evaluate vital status of patients enrolled in 3 galantamine studies | 4 weeks
  Poststudy vital status (living or deceased) of patients who participated in 3 clinical studies with galantamine will be evaluated. Data will be collected as vital status of the patient, date of death, cause of death and adverse events associated with death.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, LLC C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (144):
- United States (50):
  - Tucson, Arizona
  - Laguna Woods, California
  - Northridge, California
  - Oceanside, California
  - Paramount, California
  - San Diego, California
  - San Francisco, California
  - Hamden, Connecticut
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Fort Lauderdale, Florida
  - Miami, Florida
  - North Miami, Florida
  - Oscala F, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Paducah, Kentucky
  - Glen Burnie, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Pittsfield, Massachusetts
  - Farmington Hills, Michigan
  - Kalamazoo, Michigan
  - Clementon, New Jersey
  - Ridgewood, New Jersey
  - Summit, New Jersey
  - Albany, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - East Providence, Rhode Island
  - Providence, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Wichita Falls, Texas
  - Bennington, Vermont
  - Richmond, Virginia
  - Tacoma, Washington
  - Middleton, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Córdoba
- Australia (8):
  - Adelaide
  - Christchurch Nz
  - Hornsby Streets
  - Kew
  - Parkville
  - Perth
  - Randwick
  - Woodville
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Belgium (10):
  - Aalst
  - Antwerp
  - Hasselt
  - Jumet
  - Leuven
  - Liège
  - Merksem
  - Reet
  - Roeselare
  - Wilrijk
- Canada (21):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - North York, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Verdun, Quebec
  - Saskatoon, Saskatchewan
  - London
  - Montreal
  - North York
  - T2n
- Czechia (8):
  - Chomutov
  - Dobřany
  - Hluboká nad Vltavou
  - Kolín
  - Opava
  - Praha 8 N/A
  - Rennes Cedex
  - Ústí nad Labem
- Finland (2):
  - Helsinki
  - Kuopio
- Toulouse, France
- Germany (6):
  - Berlin
  - Frankfurt am Main
  - Mannheim
  - München
  - Nuremberg
  - Ulm
- Israel (4):
  - Haifa
  - Petach Tikya
  - Ramat Gan
  - Tel Aviv
- Netherlands (5):
  - 's-Hertogenbosch
  - Alkmaar
  - Amsterdam
  - Breda
  - Maastricht
- Poland (7):
  - Gdansk
  - Katowice Poland
  - Lodz
  - Mosina Poland
  - Poznan
  - Poznan Poland
  - Warsaw
- Spain (4):
  - Barakaldo Vizcaya S/N
  - Barcelona
  - Madrid
  - Terrasa Barcelona N/A
- Sweden (7):
  - Linköping
  - Lund
  - Malmo
  - Mölndal
  - Piteå
  - Stockholm
  - Umeå
- United Kingdom (6):
  - Bradford
  - Bristol
  - Clydebank
  - New Milton
  - Southampton
  - Swindon

REFERENCES:
- See also: Survey of the vital status of patients who participated in three studies of galantamine in treatment of mild cognitive impairment. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=573&filename=CR004240_CSR.pdf